CLINICAL TRIAL: NCT05618171
Title: Evaluation of the Patient's Pre- and Post-treatment Risk Profile Using the Peri-implantitis Risk Diagram
Brief Title: Evaluation of the Patient's Risk Profile Using the Peri-implantitis Risk Diagram
Status: Completed | Type: Observational
Sponsor: Berceste Guler (Other)
Responsible Party: Sponsor-Investigator, Berceste Guler, Associate Professor, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Other Study IDs: 2020/08-03
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Dental Implant Failed
Keywords: IDRA; Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Evaluation of the patient's pre- and post-treatment risk profile using the peri-implantitis risk diagram — By using "IDRA", a tool specially developed for patients who have had dental implants in our clinic, patients will be evaluated as "low-moderate-high" risk in terms of the risk of developing peri-implantitis, according to their initial status. Again, these patients will be re-evaluated 1 year after applying Phase I treatment using the "IDRA" tool. During this whole process, clinical and radiographic evaluations will be carried out simultaneously.

SUMMARY:
Various risk factors defined in the literature should be eliminated in order for the patient to be able to use implant-supported prostheses for a longer period of time. In the literature, such a diagram for peri-implant risk factors was first described by Heitz-Mayfield in 2020. The scheme that will determine the peri-implant risk diagram is called "Implant Disease Risk Assessment (IDRA)". This tool provides evaluation of various risk factors on a single diagram. In this study, peri-implant risk diagrams will be determined by calling the patients who have previously completed implant treatment in Kütahya University of Health Sciences Faculty of Dentistry Department of Periodontology, and the change in the risk profile assessment will be re-evaluated after the risk factors that can be eliminated are eliminated. In this study, it is aimed to predict the risk of inflammation and alveolar bone loss of the tissues around the implant that may occur in the future in patients who have undergone dental implant treatment, and to evaluate the risk profiles.

DETAILED DESCRIPTION:
Nowadays, dental implants are increasingly applied worldwide for the restoration of lost teeth. It is known that the survival rates of dental implant treatments are quite high, but in recent studies, the maintenance of the health of the peri-implant tissues and the satisfaction of the patient play a more important role in the success of the dental implant, not the survival. Various risk factors defined in the literature should be eliminated in order for the patient to be able to use implant-supported prostheses for a longer period of time. In the literature, a Spider Web scheme named "Perio-tools" has been defined, which evaluates the risk profile of the patient by determining the risk factors for periodontal diseases. However, such a diagram for peri-implant risk factors in the literature was first described by Heitz-Mayfield in 2020. The scheme that will determine the peri-implant risk diagram is called "Implant Disease Risk Assessment (IDRA)". This tool provides evaluation of various risk factors on a single diagram. In this study, peri-implant risk diagrams will be determined by calling the patients who have previously completed implant treatment in Kütahya University of Health Sciences Faculty of Dentistry Department of Periodontology, and the change in the risk profile assessment will be re-evaluated after the risk factors that can be eliminated are eliminated.

By using "IDRA", a tool specially developed for patients who have had dental implants in our clinic, patients will be grouped as "low-medium-high" risk according to their initial status in terms of the risk of developing peri-implantitis. Again, these patients will be re-evaluated using the "IDRA" tool 1 year after applying Phase I treatment. During this whole process, clinical and radiographic evaluations will be carried out simultaneously. Periapical radiographs will be taken from the implant periphery of the patients with the parallel long cone technique. According to the periodontal disease classification made in 2017, the diagnosis of the patients will be evaluated through panoramic radiographs and clinical measurements. Patients will undergo periodontal examination at their first visit. Keratinized gingival width, plaque index, gingival index, attachment loss, bleeding indices on probing will be taken. Peri-implant mucosa will be examined. Peri-implant health status will be recorded according to the following criteria.

The state of being healthy of peri-implant tissues; No bleeding on probing, no swelling, no hyperemia, no signs of inflammation Peri-implant mucositis; Inflammatory lesion limited to the soft tissues surrounding the dental implant and no bone loss Peri-implantitis; Bleeding on probing, presence of bone loss, distance between the most coronal part of the implant in the bone and the bone level ≥ 3mm, pocket depth ≥ 6mm on probing

Plaque index and gingival index are obtained by measuring 4 regions of a tooth (mesial, distal, buccal and lingual) with Williams periodontal probe.

Attachment loss: It is the value of the distance between a tooth and the free gingiva, based on the enamel-cementum junction, measured using a Williams periodontal probe.

Bleeding index in probing: In this index, probing is performed by gently walking around the pocket. As a result of probing, the evaluation is made by looking at the presence or absence of bleeding in the gingiva. If bleeding occurs within 10-15 seconds after probing in the mesial, distal, buccal and lingual gingival parts of all teeth, a positive value is given. The ratio of the bleeding area to the examined area is expressed as %.

Keratinized gingival width: It is the distance from the free gingival margin to the mucogingival junction line.

Modified plaque index and modified sulcus bleeding index will be used for implants.

Oral hygiene motivation will be given after the periodontal indexes of the patients are recorded.

If the periodontal pocket depth is excessive, routine Phase I treatment will be applied for its elimination. Likewise, risk factors related to prosthetic restoration (occlusal trauma, cement residue) will be eliminated. After all the risk factors that can be eliminated in our clinic have been eliminated, the patient will be called for a repeat risk profile evaluation 1 year later. In the follow-up of the patient 1 year later, clinical and radiographic routine evaluations will be performed again and the results will be compared.

IDRA is a functional risk assessment diagram specially developed for patients with dental implants. Evaluated data;

1. Evaluation of whether the patient has a history of periodontitis (inflammatory disease of the teeth and surrounding tissues). Studies have shown that patients with a history of periodontitis are at high risk.
2. Percentage of bleeding in periodontal probing (measurement in the gingival pocket with a periodontal probe). It has been emphasized in studies that as the percentage of bleeding on probing increases, tissue destruction increases and therefore the risk of implant loss increases.
3. Peri-implant pocket depth ≥5 mm. It is emphasized that the risk of inflammation of the tissues around the tooth and implant increases as the number of teeth or implants with a pocket depth of more than 5 mm increases.
4. Evaluation of the relationship between age and periodontal bone loss (bone loss/age). Studies emphasize that significant statistical values emerge when bone loss is compared to age.
5. Evaluation of periodontal susceptibility according to the renewed periodontal disease classification by reaching Consensus in 2017
6. Evaluation of participation in supportive periodontal therapy. Studies have emphasized the positive effects of patients' regular visits to control appointments.
7. Evaluation of the relationship between the restoration margin and the bone level. It is emphasized that the risk of inflammation of the tissues around the implant increases as the restoration margin approaches the bone crest.
8. Factors associated with dental prosthetic restoration (cleanability, evaluation of restoration compliance, etc.). It is emphasized in studies that the risk of implant loss decreases in cases where the prosthetic restorations on the implant are cleanable, well-fitted, screwed or in the absence of excessive cementation.

In this study, it is aimed to predict the risk of future inflammation of peri-implant tissues and alveolar bone loss in patients who have undergone dental implant treatment and to evaluate the risk profiles.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18
* The condition of making dental implants in Kütahya Health Sciences University, Faculty of Dentistry, Department of Periodontology
* Finding radiographic documentation of dental implants
* Functioning of the implants in the mouth for at least 1 year

Exclusion Criteria:

* Antibiotic use in the 3 months before the first examination
* Patients who have not received regular implant maintenance therapy
* Pregnant and breastfeeding women
* Mentally retarded patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent dental implants in Kütahya Health Sciences University, Faculty of Dentistry, Department of Periodontology
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of pre- and post-treatment peri-implantitis risk profiles of patients who underwent dental implant treatment at the patient level. | 1 year after phase 1 treatment
  By using "IDRA", a tool specially developed for patients who have had dental implants in our clinic, patients will be grouped as "low-medium-high" risk according to their initial status in terms of the risk of developing peri-implantitis. Again, these patients will be re-evaluated 1 year after applying Phase I treatment using the "IDRA" tool. Evaluation will be at the patient level.
Evaluation of pre- and post-treatment peri-implantitis risk profiles at implant level in patients who have undergone dental implant treatment. | 1 year after phase 1 treatment
  By using "IDRA", a tool specially developed for patients who have had dental implants in our clinic, patients will be grouped as "low-medium-high" risk according to their initial status in terms of the risk of developing peri-implantitis. Again, these patients will be re-evaluated 1 year after applying Phase I treatment using the "IDRA" tool. Evaluation will be at the implant level.

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Güler, Principal Investigator — Kütahya Health Sciences University Faculty of Dentistry
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Department of Periodontology, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It will be shared if the principal investigator is contacted.
Supporting Information: Study Protocol, CSR
Time Frame: 1 year after the research was published
Access Criteria: The principal investigator should be contacted.

REFERENCES:
- [Result] Heitz-Mayfield LJA, Heitz F, Lang NP. Implant Disease Risk Assessment IDRA-a tool for preventing peri-implant disease. Clin Oral Implants Res. 2020 Apr;31(4):397-403. doi: 10.1111/clr.13585. Epub 2020 Feb 20. PMID 32003037
- [Result] Dalago HR, Schuldt Filho G, Rodrigues MA, Renvert S, Bianchini MA. Risk indicators for Peri-implantitis. A cross-sectional study with 916 implants. Clin Oral Implants Res. 2017 Feb;28(2):144-150. doi: 10.1111/clr.12772. Epub 2016 Jan 11. PMID 26754342